CLINICAL TRIAL: NCT07156513
Title: Pulsed Epidural Radiofrequency Versus Epidural Steroid Injection in Patients With Failed Back Syndrome
Brief Title: Persistent Post-Lumbar Surgery Pain Syndrome (PSPS) Type II is a Common Condition Encountered in Pain Units, With Limited Available Therapeutic Options. Epidural Pulsed Radiofrequency (PRF) Administered Via Catheter Has Demonstrated Greater Efficacy Compared to the Transforaminal Approach. This Rand
Acronym: EPIPUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Agustin Mendiola de la Osa, MD, PhD, MBA, FIPP, CIPS, EDPM, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Epipul Study; Comité Ético de HM Hospital (Other: Código CEIm HM Hospitales: 20.07.1662-GHM)
Record Dates: First submitted 2025-08-13; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Persistent Spinal Pain Syndrome Type II; Failed Back Surgery Syndrome; Chronic Low Back Pain; Post-Laminectomy Syndrome
Keywords: PRF Catheter; Epidural Steroid Injection; Neuropathic Pain; Interventional Pain Management; Epidural Pulsed Radiofrequency
MeSH Terms: conditions — Failed Back Surgery Syndrome; post laminectomy syndrome; Neuralgia | interventions — Betamethasone

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, multicenter, parallel-group study. Participants were assigned in a 1:1 ratio to receive either epidural corticosteroid injection alone (control group) or epidural pulsed radiofrequency combined with corticosteroid injection (experimental group).
Who Masked: Participant
Masking Description: Participants were blinded to treatment assignment. Care providers and investigators were aware of group allocation in order to perform the procedures. No additional parties were masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Arm (Experimental): Participants received epidural pulsed radiofrequency with corticosteroid injection.
  Interventions: Procedure: Epidural Pulsed Radiofrequency; Drug: Betamethasone (Epidural Corticosteroid Injection)
- Control Arm: Epidural Corticosteroid Injection (Active Comparator): Participants received an epidural injection of 12 mg betamethasone in 8 ml sterile saline without pulsed radiofrequency.
  Interventions: Drug: Betamethasone (Epidural Corticosteroid Injection)

INTERVENTIONS:
Procedure: Epidural Pulsed Radiofrequency — Pulsed radiofrequency applied via a guidable epidural catheter electrode (Cosman RCE-E401519-P), advanced through the sacral hiatus to the target lumbar or sacral root (L5 and/or S1) under fluoroscopic guidance. Parameters: 45 V, 2 Hz, 20 ms pulses, applied at a single location with continuous temperature monitoring (≤42°C). Procedure performed with Cosman C4 generator.
  Arms: Experimental Arm
Drug: Betamethasone (Epidural Corticosteroid Injection) — Epidural injection of 12 mg betamethasone diluted in 8 ml sterile saline, administered via the sacral hiatus under fluoroscopic guidance.

SUMMARY:
This study is for people who continue to have low back pain after spinal surgery, a condition called persistent spinal pain syndrome type II. Current treatments, such as epidural injections, often provide only limited relief. Doctors are testing a procedure called pulsed radiofrequency (PRF), given through a small catheter in the epidural space, with or without the addition of corticosteroids. The goal is to see if this treatment can reduce pain and improve daily function better than standard injections. About 130 patients took part, and their pain and quality of life were followed for several months after the procedure.

DETAILED DESCRIPTION:
Persistent spinal pain syndrome type II (PSPS II) is a frequent and disabling condition encountered in Pain Units after lumbar surgery. Conventional therapeutic options such as epidural corticosteroid injections and epidurolysis often provide only partial or temporary benefit. Pulsed radiofrequency (PRF) delivered through a catheter into the epidural space has shown promising results compared to transforaminal approaches, offering a potential alternative for managing this challenging pain condition.

The purpose of this randomized, controlled, multicenter clinical trial is to evaluate the efficacy and safety of epidural PRF with or without the addition of corticosteroids in patients with PSPS II. A total of 131 patients were enrolled and assigned to receive either epidural corticosteroids alone or PRF combined with corticosteroids. Pain intensity, functional status, neuropathic pain features, and global impression of improvement were assessed at multiple follow-up visits. The findings of this study aim to provide evidence-based guidance for interventional pain management in PSPS II.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years old.
2. Written informed consent obtained according to ICH/GCP and Spanish legislation prior to any study procedure.
3. Pain VAS score of at least 5 points.
4. Duration of pain lasting at least 3 months after back surgery despite conservative treatment.
5. Leg-dominant radicular pain deemed neuropathic based on clinical history and examination.
6. Responsiveness to selective radicular nerve block with bupivacaine 0.125%.
7. Previous epidural steroid injection.

Exclusion Criteria:

1. Pregnancy or lactation. 2. Participation in a study involving medicines or other clinical devices 4. Inability to follow instructions or collaborate during the study. 5. Findings in physical examination, clinical analysis abnormalities, or other medical, social, or psychosocial factors that, in the researcher's opinion, could negatively influence study outcomes 6. Presence of myelopathy, systemic diseases, infection (systemic or local), cancer, indication for immediate surgery, coagulation disorders, anticoagulants use, diabetes mellitus or multiple sclerosis.

7. Life expectancy of less than one year. 8. Current diagnosis of a progressive neurological disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity measured by Visual Analogue Scale (VAS) | Baseline to 6 months (with assessments at 1, 2, 4, and 6 months).
  Change in pain intensity measured by the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in neuropathic pain measured by DN4 questionnaireeuropathic pain, as measured by DN4 questionnaire | Time Frame: Baseline to 6 months (assessments at 1, 2, 4, and 6 months).
  Description: Neuropathic pain assessed using the Douleur Neuropathique 4 Questions (DN4), with scores ranging from 0 to 10. Higher scores indicate greater neuropathic pain.
Change in functional disability measured by Oswestry Disability Index (ODI) | Baseline to 6 months (assessments at 1, 2, 4, and 6 months)
  Description: Functional disability assessed using the Oswestry Disability Index (ODI), with scores ranging from 0% (no disability) to 100% (maximum disability).
Change in overall improvement measured by Patient Global Impression of Improvement (PGI-I) questionnaire | Baseline to 6 months (assessments at 1, 2, 4, and 6 months).
  Description: Overall patient improvement assessed using the Patient Global Impression of Improvement (PGI-I) scale, ranging from 1 (very much improved) to 7 (very much worse).

OTHER OUTCOMES:
Number Needed to Treat (NNT) analysis for pain reduction | Baseline to 6 months (assessments at 1, 2, 4, and 6 months).
  Description: Number Needed to Treat (NNT) will be calculated based on the proportion of patients achieving clinically relevant reductions in pain intensity on the VAS (e.g., ≥2-point or ≥3-point reduction). Lower NNT values indicate greater treatment efficacy

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - HM Monteprincipe University Hospital, Boadilla del Monte, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - General Hospital Of Ciudad Real, Ciudad Real
  - HM Sanchinarro University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this article will be available upon reasonable request to the Principal Investigator (Dr. Agustín Mendiola de la Osa) after publication. Data will be shared for research purposes only, following approval of a methodologically sound proposal and under a data access agreement.
Supporting Information: SAP, ICF, CSR
Time Frame: Data will be available from the publication date of the main results and for 5 years thereafter.
Access Criteria: De-identified IPD, including baseline data, intervention details, and outcomes (VAS, ODI, DN4, PGI-I), will be available to qualified researchers upon reasonable request. Proposals require approval by the principal investigator and ethics committee. Access will be granted after signing a data use agreement and will be provided via secure electronic transfer.
URL: https://1drv.ms/w/c/66ca2196fe0a03bd/Ed0zlbWharVCpK2AmmPOAFMB1umlwjzN2JKMM9vmF_4CDg

REFERENCES:
- [Background] Chua NH, Vissers KC, Sluijter ME. Pulsed radiofrequency treatment in interventional pain management: mechanisms and potential indications-a review. Acta Neurochir (Wien). 2011 Apr;153(4):763-71. doi: 10.1007/s00701-010-0881-5. Epub 2010 Nov 30. PMID 21116663
- [Background] Gulduren Aydin LG, Akesen S, Turker YG, Gurbet A, Kilic Yilmaz V. Investigation of Effectiveness of Pulsed Radiofrequency With Multifunctional Epidural Electrode for Low Back Pain. Cureus. 2021 Dec 7;13(12):e20239. doi: 10.7759/cureus.20239. eCollection 2021 Dec. PMID 35004054
- [Background] Abejon D, Garcia-del-Valle S, Fuentes ML, Gomez-Arnau JI, Reig E, van Zundert J. Pulsed radiofrequency in lumbar radicular pain: clinical effects in various etiological groups. Pain Pract. 2007 Mar;7(1):21-6. doi: 10.1111/j.1533-2500.2007.00105.x. PMID 17305674
- [Background] Petersen EA, Schatman ME, Sayed D, Deer T. Persistent Spinal Pain Syndrome: New Terminology for a New Era. J Pain Res. 2021 Jun 8;14:1627-1630. doi: 10.2147/JPR.S320923. eCollection 2021. No abstract available. PMID 34135626

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT07156513/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT07156513/ICF_001.pdf